CLINICAL TRIAL: NCT03415269
Title: A Single-Centre, Open-label, Exploratory Study of the Effect of 20 mg Ambroxol Hydrochloride on Cough Reflex Sensitivity in Patients With Acute Cough.
Brief Title: A Study of the Effect of 20 mg Ambroxol Hydrochloride on Acute Cough.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIT15419
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2018-01

CONDITIONS: Cough
Keywords: acute
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 mg ambroxol (Experimental): 20 mg ambroxol lozenge delivered once on one day
  Interventions: Drug: Ambroxol Hydrochloride

INTERVENTIONS:
Drug: Ambroxol Hydrochloride — single lozenge of 20mg ambroxol
  Other Names: Lysopain Ambr Mint™

SUMMARY:
To assess the effect of a single doses of 20 mg ambroxol hydrochloride on cough reflex sensitivity to citric acid, capsaicin, adenosine triphosphate (ATP) and distilled water in patients with acute cough related to upper respiratory tract infection

DETAILED DESCRIPTION:
Cough is the 5th most common presenting complaint in adults. Cough results from the stimulation of two types of afferent pathways whose receptors are located within the airway epithelium. These include rapidly adapting receptors (RARs) and C-fibre receptors. Acute as well as chronic, non-productive cough, which often follow viral upper respiratory tract infection, may result from increased sensitivity of the cough reflex. Relatively little research has been done to gain insight into the mechanisms of cough in health and disease, and to properly evaluate potential antitussive therapies. Indeed, little consensus exists regarding the optimal treatment of acute cough because of the lack of standardised outcome measures for cough. Possibly the most significant clinical need in terms of cough therapy is for the cough associated with an acute upper respiratory tract infection (URTI). Although the cough associated with URTI is often self-limiting and resolves within several days, it undoubtedly accounts for a major proportion of huge worldwide expenditure of over-the-counter (OTC) cough and cold products where patients are still struggling to find an effective medication.

This exploratory study will enable us to identify the cough challenge agent (CCA) that is most sensitive to the effect of ambroxol on cough reflex. This is expected to provide a reproducible response, to use in future studies.

This will be an open label, study in subjects with acute cough associated with URTI.

There will be a Screening/Baseline and combined Treatment visit. Subjects will return approximately 1-4 weeks after their treatment once all symptoms have subsided and the subject is no longer suffering from URTI, for a Follow-up Visit.

Up to 14 subjects with acute cough in relation to a URTI and who meet all entry criteria will be assigned to:

Treatment p.o 20 mg ambroxol lozenge (Lysopain Ambr MintM)

At Baseline and post treatment, cough sensitivity will be measured by standard clinical methodology incorporating a series of four cough challenges (citric acid, capsaicin, ATP and distilled water).

Screening/baseline visit 1a The Screening and Baseline visit will ensure that each subject meets all the specified inclusion and none of the exclusion criteria.

Treatment phase visit 1b Subjects who satisfy all entry criteria at baseline will be administered 20 mg ambroxol in the form of a lozenge which must be sucked until fully dissolved in the mouth.

The treatment will be administered in the afternoon of the same visit day as the screening/baseline assessments.

The series of abbreviated cough challenges will be conducted at 30 min and 90 min post dose.

Telephone contact Patients will be contacted by telephone once a week to determine if all symptoms associated with URTI have abated. Once this is confirmed patient will be booked in for the follow-up visit.

Follow-Up Phase Subjects will return within 4 weeks after treatment for a Follow-Up Visit once symptoms of URTI have abated. A series of full cough challenges will be performed at this vist to determine reduction in cough hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed of the nature of the study and have provided written informed voluntary consent;
2. Be able to speak, read, and understand English;
3. Be males or females, of any race, between 18 and 80 years of age, inclusive;
4. Subject has an acute cough and other symptoms consistent with a common cold or an acute upper respiratory tract infection (URTI) diagnosis deemed by the investigator based on findings from medical history review, full physical examination and vital signs;
5. The onset of symptoms must be within 72 h of study enrolment;
6. Have a Cough Severity VAS ≥ 40 mm at Screening;
7. Be in good general health (other than URTI) with no clinically relevant abnormalities based on the medical history, physical examination, and 12 lead electrocardiogram;
8. Cough at least twice to all cough challenge Agents - citric acid, capsaicin, ATP and distilled water cough challenges at baseline.
9. If a female of child-bearing potential (i.e., have not undergone a hysterectomy or bilateral oophorectomy) or not post-menopausal (defined as no menses for at least 12 months), agree to use 2 forms of acceptable birth control from Screening through to the Follow Up Visit; or if a male, they and/or their partner of child-bearing potential agree to use 2 forms of acceptable birth control from Screening through the Follow Up Visit;
10. Be able to communicate effectively with the Investigator and other study centre personnel and agree to comply with the study procedures and restrictions.

    -

    Exclusion Criteria:
11. History of asthma or other respiratory related disease
12. Symptoms of runny nose, stuffy nose, sore throat, or sneezing due to any condition other than URTI or common cold (e.g., seasonal or perennial allergic rhinitis, sinusitis, strep throat, vasomotor rhinitis, etc.) as established by the investigator
13. Clinical features of a complication of the common cold during the physical examination at screening (e.g., otitis media, sinusitis, or pneumonia) with or without the need for systemic antibiotics
14. History of a severe cutaneous adverse reaction to any treatment;
15. Evidence of a possible bacterial infection i.e. sinus pain, purulent nasal discharge or pleuritic pain.
16. Evidence of chest infection or pneumonia
17. Fever greater than 39ºC (102ºF oral temperature) at the time of screening if, in the judgment of the investigator, the individual is too ill to participate in the study or the fever is due to reasons other than URTI
18. Demonstrate more than two coughs to inhalation of the normal saline solution during baseline challenge
19. Current smoker or individuals who have given up smoking within the past 6 months or those with >20 pack-year smoking history;
20. Treatment with an ACE-inhibitor during the study or within 4 weeks prior to Screening
21. History of opioid use within 1 week prior to baseline;
22. Requiring concomitant therapy with prohibited medications
23. History of known or suspected allergy or hypersensitivity reactions to ambroxol (e.g., asthma, urticaria or allergic type) or any of the non-medicinal ingredients contained in the study investigational product.
24. Clinically significant abnormal electrocardiogram (ECG) at Screening;
25. Personal or family history of congenital long QT syndrome or family history of sudden death;
26. Pregnant or breastfeeding;
27. Treatment with an investigational drug or biologic within 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion;
28. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the subject inappropriate for entry into this trial -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Cough reflex sensitivity | 8 hours
  To assess the effect of single dose of 20 mg ambroxol lozenge on cough reflex sensitivity (quatified by recording the concenteration of cough stimulant evoking 2 (C2) and 5 (C5 ) coughs) to four different types of challenge agents in acute cough associated with URTI.

SECONDARY OUTCOMES:
Severity of cough Visual analogue scale (VAS) | 90 min post dose
  To determine the effect of single dose of 20 mg ambroxol lozenge on cough severity Visual analogue Scale from baseline compared to 30 min and 90 min post ambroxol 20 mg. The visual analogue scale will comprise of a 100mm horizontal line representing a scale of cough severity from 'No Cough' at the left hand (0 mm) end of the line up to 'Worst Cough'(100mm) at the right hand end. The participant will be instructed to draw a single vertical line on the scale to indicate how severe they felt their cough has been during a specified time.
Urge to cough Visual analogue scale (VAS) | 90 min post dose
  To determine the effect of single dose of 20 mg ambroxol lozenge on urge to cough VAS from baseline compared to 30 min and 90 min post ambroxol 20 mg The Visual analogue scale will be a 100mm scale used to record the severity of their urge to cough but marked at the extremes as 'No urge-to-cough' on the left side (0mm) and 'Worst urge-to-cough' (100 mm) on the right side. The participant is instructed to draw a single vertical line on the scale to indicate how severe their urge to cough was during a specified time.
Change in cough reflex sensitivity from during acute cough to post symptom recovery | up tp 1 month
  measure change in cough reflex sensitivity to citric acid, capsaicin, ATP and distilled water as measured using the C2 and C5 and compare this to that measured post symptom recovery

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03415269/SAP_000.pdf